CLINICAL TRIAL: NCT00159822
Title: Voriconazole For Primary Therapy Of Proven, Chronic Bronchopulmonary Aspergillosis, In Minimally Immunocompromised Or, Non-Immunocompromised Hosts
Brief Title: Voriconazole For Chronic Bronchopulmonary Aspergillosis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A1501061
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Results first posted 2010-01-07 (Estimated); Last update posted 2010-01-20 (Estimated); Status verified 2010-01

CONDITIONS: Aspergillosis
MeSH Terms: conditions — Aspergillosis | interventions — Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Voriconazole

INTERVENTIONS:
Drug: Voriconazole — Voriconazole oral : loading dose on day 1 : 400mg/12 hours; maintenance dose 200 mg /12 hours for 6 to 12 months depending on clinical response.
  Alternatively, patients may start on Voriconazole, IV, for 7 days loading dose, 6mg/Kg/12 hours on day one and maintenance dose 4 mg/Kg/12 hours

SUMMARY:
To evaluate the efficacy of voriconazole (VFend(R)) as first line treatment for proven chronic bronchopulmonary aspergillosis, in minimally immunocompromised or non-immunocompromised patients after 6 months of treatment i.e. chronic necrotizing pulmonary

ELIGIBILITY:
Inclusion Criteria:

* Patients with a chronic bronchopulmonary aspergillosis assessed by a compatible chest imagery (CT scan) and/or an endoscopic lesion sourced by photo, would it be:
* Complex aspergilloma non primarily operable,
* Chronic necrotizing pulmonary aspergillosis,
* Tracheo-bronchial aspergillosis, obstructive or necrotizing/pseudo-membranous.

Exclusion Criteria:

* Patient with risk factor(s) of cardiac arrhythmia, symptomatic arrhythmia, treated by medication known to prolong QT interval, or prolongation of QTc interval > 450 msec in men and > 470 msec in women.
* Simple aspergilloma with primary indication of surgical treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-07; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (16):
- France (16):
  - Pfizer Investigational Site, Nantes, Cedex
  - Pfizer Investigational Site, Angers
  - Pfizer Investigational Site, Bobigny
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Bris Sous Forges
  - Pfizer Investigational Site, Caen
  - Pfizer Investigational Site, Dinan
  - Pfizer Investigational Site, Grenoble
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Poitiers
  - Pfizer Investigational Site, Reims
  - Pfizer Investigational Site, Rouen
  - Pfizer Investigational Site, Suresnes

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1501061&StudyName=Voriconazole%20and%20Bronchopulmonary%20Aspergillosis%20

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 18 active centers in France; planned recruitment of 48 minimally immunocompromised or non-immunocompromised subjects with chronic bronchopulmonary aspergillosis.
Pre-assignment Details: 56 subjects were screened; 48 subjects included; 8 subjects did not meet criteria and were not included.
Groups:
- Voriconazole: Voriconazole (VFend®) initially administered intravenously (IV) or orally (PO) based on investigator's clinical decision. PO loading dose every 12 hours on Day 1 for body weight ≥ 40 kilograms (kg): 400 milligrams (mg) followed by maintenance dose of 200 mg every 12 hours; or for body weight < 40 kg, loading dose every 12 hours on Day 1: 200 mg followed by maintenance dose of 100 mg every 12 hours. If initially IV, loading dose every 12 hours on Day 1: 6 mg/kg followed by maintenance dose of 4 mg/kg every 12 hours for 3 to 10 days; then, switched to PO maintenance dose based on body weight.
Period: Voriconazole Treatment Period
Arm/Group | Voriconazole
Started | 48
Completed | 26 (Number of subjects completed treatment: 36 up to month 6 (M6); 26 after M6.)
Not Completed | 22
Not completed — Lack of Efficacy | 3
Not completed — Adverse Event | 9
Not completed — Death | 4
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 2
Period: Post-treatment Follow-up Period
Arm/Group | Voriconazole
Started | 26
Completed | 23
Not Completed | 3
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Reason unspecified | 1

BASELINE CHARACTERISTICS:
Arm/Group | Voriconazole
Number analyzed (Participants) | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 57.27 (13.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Successful Global Outcome at 6 Months: Chronic Bronchopulmonary Aspergillosis
Description: Successful global outcome: composite assessment of radiological and mycological responses; defined as complete or partial radiological response and mycological eradication (absence of aspergillus); no success=criteria not met. Assessment was determined by the Data Review Committee (DRC). Complete response: resolution of radiographic and or bronchoscopic abnormalities attributable to aspergillosis present at baseline; partial response: reduction in diameter ≥ 50 percent on chest tomodensitometry (TDM) or regressed lesion on endoscopy witnessed by 2 different operators without any new lesion.
Time Frame: at 6 months of treatment
Population: Modified Intent to Treat (mITT): all subjects in ITT population (took at least 1 dose of voriconazole and had at least 1 post-inclusion efficacy assessment) who had diagnosis of chronic bronchopulmonary aspergillosis confirmed by the Data Review Committee (DRC); 5 subjects excluded from mITT population due to unproven diagnosis.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 41
participants
  Success | 13
  No success | 28
Statistical Analysis 1: Comparison: Voriconazole; For sample size calculation, null hypothesis (p<p0) is defined as response rate <15% (ie, weak drug efficacy). Alternative hypothesis (p>pA) defined as response rate >30%. To reduce the chance of incorrectly rejecting the null hypothesis to 5% (α=5%) and incorrectly rejecting the alternate hypothesis to 20% (β=20%) it was calculated that a sample size of 48 subjects was required. Null hypothesis was rejected (assessing efficacy of study drug) if the number of eligible success was ≥ than n=12; Test type: Superiority or Other; Percent of subjects with success = 31.7, 95% CI [18.08 to 48.09] — Number of subjects with successful global outcomes were summarized and 95% two-sided confidence intervals based on the exact Clopper-Pearson method for the binomial distribution provided

2. Secondary Outcome: Number of Subjects With Successful Global Outcome at Month 3 and End of Treatment: Chronic Bronchopulmonary Aspergillosis
Description: Successful global outcome: composite assessment of radiological and mycological responses; defined as complete (resolution of radiographic and or bronchoscopic abnormalities attributable to aspergillosis present at baseline) or partial (reduction in diameter ≥ 50 percent on chest TDM or regressed lesion on endoscopy witnessed by 2 different operators without any new lesion) radiological response and mycological eradication after 3 months of treatment and after 9 or 12 months (in case of extension of treatment period beyond 6 months); no success=criteria not met. Assessment determined by DRC.
Time Frame: Month 3 and End of Treatment (Month 9 or Month 12)
Population: mITT; End of treatment (EOT) or at last visit available [LVA] (EOT or LVA includes data from 6, 9 or 12 months in case of extension of the treatment period beyond 6 months). Month 6 analysis is reported in the primary outcome measure.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 41
participants
  Month 3 success=yes | 12
  Month 3 success=no | 24
  Month 3 success=missing values | 5
  EOT [LVA] success=yes | 18
  EOT [LVA] success=no | 23
Statistical Analysis 1: Comparison: Voriconazole; Month 3 success=yes; Test type: Superiority or Other; Percent of subjects with success = 33.3, 95% CI [18.6 to 51.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Voriconazole; EOT success=yes; Test type: Superiority or Other; Percent of subjects with success = 43.9, 95% CI [28.5 to 60.3] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Number of Subjects With Successful Global Outcome at 6 Months: Chronic Necrotizing Pulmonary Aspergillosis (CNPA) and Tracheo-bronchial Aspergillosis
Description: Successful global outcome: composite assessment of radiological and mycological responses; defined as complete or partial radiological response and mycological eradication (absence of aspergillus); no success=criteria not met. Assessment was determined by the Data Review Committee (DRC). Complete response: resolution of all radiographic and or bronchoscopic abnormalities attributable to the aspergillosis present at baseline; partial response: reduction in diameter ≥ 50% on chest tomodensitometry (TDM) or regressed lesion on endoscopy witnessed by 2 different operators without any new lesion.
Time Frame: at 6 months of treatment
Population: mITT
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 19
participants
  Success | 10
  No success | 9

4. Secondary Outcome: Number of Subjects With Successful Global Outcome at 6 Months: Complex Aspergilloma
Description: as for outcome 3
Time Frame: at 6 months of treatment
Population: mITT
Measure: Number; unit: paticipants
Arm/Group | Voriconazole
Number analyzed (Participants) | 22
paticipants
  Success | 3
  No success | 19

5. Secondary Outcome: Change From Baseline in Respiratory Clinical Signs and Symptoms on Visual Analog Scales (VAS)
Description: Subject assessment of improvement of respiratory clinical signs and symptoms as indicated by the subject placing a mark on a 10 cm VAS scored 0 (better state of health) to 100 (poor state of health) for cough, dyspnea, sputum, hemoptysis, chest tightness, and nocturnal awakening. Change from baseline: mean of (value of scores on scale at treatment visit minus baseline value).
Time Frame: Baseline, Month 3, and Month 6, Month 9, or Month 12 [EOT], and End of study ([EOS] EOT + 6 months)
Population: mITT; 6, 9 or 12 months (in case of extension of the treatment period beyond 6 months) as EOT or last visit available; (n) = number of subjects with analyzable data at observation. Subject may be represented in >1 category.
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Voriconazole
Number analyzed (Participants) | 41
scores on scale
  Cough Month 3 (n=30) | -15.80 (33.40) [-28.27 to -3.33]
  Cough Month 6 (n=27) | -19.63 (35.48) [-33.67 to -5.59]
  Cough Month 9 (n=20) | -17.45 (43.01) [-37.58 to 2.68]
  Cough Month 12 (n=16) | -30.13 (37.01) [-49.85 to -10.40]
  Cough EOS (n=20) | -13.65 (41.31) [-32.98 to 5.68]
  Dyspnea Month 3 (n=30) | -2.67 (24.22) [-11.71 to 6.38]
  Dyspnea Month 6 (n=27) | -4.22 (25.16) [-14.17 to 5.73]
  Dyspnea Month 9 (n=20) | -1.40 (24.66) [-12.94 to 10.14]
  Dyspnea Month 12 (n=16) | -8.69 (25.15) [-22.09 to 4.71]
  Dyspnea EOS (n=20) | 1.75 (31.30) [-12.90 to 16.40]
  Sputum Month 3 (n=30) | -8.03 (27.44) [-18.28 to 2.21]
  Sputum Month 6 (n=28) | -14.86 (37.11) [-29.25 to -0.47]
  Sputum Month 9 (n=21) | -12.62 (37.35) [-29.62 to 4.38]
  Sputum Month 12 (n=17) | -26.47 (26.59) [-40.14 to -12.80]
  Sputum EOS (n=21) | -13.67 (36.20) [-30.15 to 2.81]
  Hemoptysis Month 3 (n=30) | -2.13 (28.05) [-12.61 to 8.34]
  Hemoptysis Month 6 (n=28) | 5.11 (27.41) [-5.52 to 15.73]
  Hemoptysis Month 9 (n=21) | -4.52 (30.32) [-18.33 to 9.28]
  Hemoptysis Month 12 (n=16) | -8.31 (31.44) [-25.07 to 8.44]
  Hemoptysis EOS (n=21) | 1.14 (20.72) [-7.73 to 10.02]
  Chest tightness Month 3 (n=30) | 0.03 (37.85) [-14.10 to 14.17]
  Chest tightness Month 6 (n=28) | 0.86 (29.83) [-10.71 to 12.42]
  Chest tightness Month 9 (n=21) | -1.52 (33.03) [-16.56 to 13.51]
  Chest tightness Month 12 (n=17) | -9.29 (31.27) [-25.37 to 6.78]
  Chest tightness EOS (n=20) | -4.00 (22.31) [-14.44 to 6.44]
  Nocturnal awakening Month 3 (n=30) | 0.57 (29.33) [-10.39 to 11.52]
  Nocturnal awakening Month 6 (n=28) | -2.86 (36.84) [-17.14 to 11.43]
  Nocturnal awakening Month 9 (n=21) | -2.40 (31.13) [-16.57 to 11.76]
  Nocturnal awakening Month 12 (n=16) | 4.00 (31.45) [-12.76 to 20.76]
  Nocturnal awakening EOS (n=21) | 5.29 (41.96) [-13.81 to 24.38]
  Mean VAS Month 3 (n=30) | -4.67 (18.29) [-11.50 to 2.16]
  Mean VAS Month 6 (n=27) | -5.99 (20.82) [-14.22 to 2.25]
  Mean VAS Month 9 (n=20) | -7.16 (24.31) [-18.54 to 4.21]
  Mean VAS Month 12 (n=15) | -15.87 (20.67) [-27.32 to -4.42]
  Mean VAS EOS (n=19) | -6.58 (20.43) [-16.43 to 3.27]

6. Secondary Outcome: Number of Subjects With Relapse
Description: Relapse: any proven reappearance of pulmonary aspergillosis during the follow-up period, following a successful global outcome at EOT, and defined as a deterioration of clinical signs and symptoms, confirmed radiologically (chest [TDM] and or endoscopy) and mycologically (histology and or culture and or serology).
Time Frame: During the 6 months following EOT (EOT + 3 months, EOT + 6 months)
Population: mITT; due to the small number of radiological reappearance (4 subjects), no formal analysis of this endpoint was performed.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 0

7. Secondary Outcome: Time to Relapse After EOT
Description: Time (months) to relapse: any proven reappearance of pulmonary aspergillosis during the follow-up period, following a successful global outcome at EOT, and defined as a deterioration of clinical signs and symptoms, confirmed radiologically (chest [TDM] and or endoscopy) and mycologically (histology and or culture and or serology).
Time Frame: During the 6 months following EOT (EOT + 3 months, EOT + 6 months)
Population: as for outcome 6
Measure: Number; unit: months
Arm/Group | Voriconazole
Number analyzed (Participants) | 0

8. Secondary Outcome: Global Survival: Number of Subjects With an Outcome of Death
Description: Number of subjects with an outcome of death (adverse event with a fatal outcome) through end of study.
Time Frame: Baseline through EOS (EOT + 6 months)
Population: Safety population (SAF): all subjects who took at least 1 dose of voriconazole.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 48
participants | 5 [0.725 to 0.976]
Statistical Analysis 1: Comparison: Voriconazole; Test type: Superiority or Other; Kaplan-Meier estimate overall survival = 0.850, 95% CI [0.725 to 0.976] — Global survival rate calculated using Kaplan-Meier estimate of overall survival

9. Secondary Outcome: Change From Baseline in Quality of Life (QOL): St. George's Hospital Respiratory Questionnaire
Description: Subject administered questionnaire to measure improvement in QOL; 50 questions exploring 3 different areas: symptoms, impact on activity profile (activity), and impact on daily life (impacts). Each item in an area is weighted based on empirical data; scores range from lowest possible weight 0 to highest possible weight 100. Scores for each section and total score calculated using score calculation algorithms with higher scores indicating poor health. Change from baseline: mean of (value of scores on scale at treatment visit minus baseline value).
Time Frame: Baseline, Month 3, and Month 6, Month 9, or Month 12 [EOT], and EOS (EOT + 6 months)
Population: mITT; 6, 9 or 12 months (in case of extension of the treatment period beyond 6 months) as EOT or last visit available; (n) = number of subjects with analyzable data at observation.
Measure: Mean (95% Confidence Interval); unit: scores on scale
Arm/Group | Voriconazole
Number analyzed (Participants) | 41
scores on scale
  Symptoms Month 3 (n=35) | -5.50 (22.53) [-13.24 to 2.24]
  Symptoms Month 6 (n=29) | -3.32 (7.37) [-14.01 to 7.37]
  Symptoms Month 9 (n=19) | 0.96 (29.78) [-13.39 to 15.32]
  Symptoms Month 12 (n=17) | -2.72 (23.80) [-14.95 to 9.52]
  Symptoms EOS (n=23) | -6.84 (23.53) [-17.01 to 3.34]
  Activity Month 3 (n=31) | -4.15 (17.72) [-10.65 to 2.35]
  Activity Month 6 (n=28) | -9.43 (17.30) [-16.13 to -2.72]
  Activity Month 9 (n=18) | -0.03 (18.04) [-9.00 to 8.94]
  Activity Month 12 (n=18) | -5.88 [-10.98 to -0.78]
  Activity EOS (n=23) | -8.06 [-14.58 to -1.54]
  Impacts Month 3 (n=33) | -6.72 [-12.42 to -1.03]
  Impacts Month 6 (n=28) | -8.41 [-15.22 to -1.61]
  Impacts Month 9 (n=20) | -3.78 [-14.72 to 7.16]
  Impacts Month 12 (n=18) | -7.97 [-16.49 to 0.55]
  Impacts EOS (n=21) | -7.93 [-13.46 to -2.40]
  Total Month 3 (n=35) | -5.70 [-10.60 to -0.81]
  Total Month 6 (n=30) | -8.39 [-14.02 to -2.76]
  Total Month 9 (n=20) | -1.87 [-11.26 to 7.51]
  Total Month 12 (n=18) | -6.63 [-12.97 to -0.28]
  Total EOS (n=24) | -8.19 [-12.41 to -3.96]

10. Secondary Outcome: Number of Subjects With Complete or Partial Radiological Response
Description: Radiological response: based on chest TDM except for tracheo-bronchialaspergillosis which was assessed by bronchoscopy. Complete response: resolution of all radiographic and or bronchoscopic abnormalities attributable to aspergillosis present at baseline; partial response: reduction in diameter ≥ 50% on chest TDM or regressed lesion on endoscopy witnessed by 2 different operators without any new lesion.
Time Frame: Month 3, and Month 6, Month 9, or Month 12 [EOT]
Population: mITT; End of treatment (EOT) or at last visit available [LVA](EOT or LVA includes data from 6, 9 or 12 months in case of extension of the treatment period beyond 6 months).
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 37
participants
  Month 3 Complete response | 4
  Month 3 Partial response | 9
  EOT [LVA] Complete response | 6
  EOT [LVA] Partial response | 14

11. Secondary Outcome: Number of Subjects With Mycological Response of Eradication
Description: Mycological response: eradication: absence of aspergillus species (spp) in bronchopulmonary samples: sputum, bronchial aspirate or bronchoalveolar lavage (BAL) (negative direct examination [exam] and negative culture), and negative histological exam when available; persistence (no eradication): presence of aspergillus spp in any relevant bronchopulmonary samples. Not done (presumed eradication): case reviewed by DRC for any mycological exams not performed to assess if case should constitute presumed eradication (no sputum due to clinical improvement).
Time Frame: Month 3, and Month 6, Month 9, or Month 12 [EOT]
Population: mITT; 6, 9 or 12 months (in case of extension of the treatment period beyond 6 months) as EOT or last visit available.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 35
participants
  Month 3 Eradication | 29
  Month 3 Persistence | 3
  Month 3 Not done (presume eradication) | 3
  Month 6 Eradication | 26
  Month 6 Not done (presume eradication) | 6
  Month 9 Eradication | 14
  Month 9 Not done (presume eradication) | 7
  Month 12 Eradication | 15
  Month 12 Not done (presume eradication) | 2

12. Secondary Outcome: Number of Subjects With Complete or Partial Serological Response
Description: Serological response: normalization (complete response) defined as return to normal values (≤ 1 arc); partial response defined as significant decrease but not complete (decrease of 2 or more arcs compared to baseline). Complete or partial response summarized as Improvement; based on arc values at visit compared to arc values at baseline (inclusion).
Time Frame: Month 3, and Month 6, Month 9, or Month 12 [EOT]
Population: mITT (with serology at inclusion); 6, 9 or 12 months (in case of extension of the treatment period beyond 6 months) as EOT or last visit available. Data summarized as Worsening (failure), No change (stabilization), or Improvement (complete or partial response) due to large number of missing results values.
Measure: Number; unit: participants
Arm/Group | Voriconazole
Number analyzed (Participants) | 40
participants
  Month 3 Improvement | 10
  Month 6 Improvement | 14
  Month 9 Improvement | 9
  Month 12 Improvement | 8

ADVERSE EVENTS:
Description: Safety population (SAF): consisted of all subjects who took at least one dose of voriconazole.
Arm/Group | Voriconazole
Serious Adverse Events (participants affected / at risk) | 21/48
Other Adverse Events (participants affected / at risk) | 33/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole (N=48)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
General physical health deterioration (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Bronchitis (Infections and infestations) | 2
Bronchitis haemophilus (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pseudomonas bronchitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
General physical condition abnormal (Investigations) | 1
Weight decreased (Investigations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary pneumatocele (Respiratory, thoracic and mediastinal disorders) | 1
Arterial stent insertion (Surgical and medical procedures) | 1
Surgery (Surgical and medical procedures) | 1
Peripheral ischaemia (Vascular disorders) | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Voriconazole (N=48)
Vision blurred (Eye disorders) | 6
Visual impairment (Eye disorders) | 9
Constipation (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Vomiting (Gastrointestinal disorders) | 3
Chills (General disorders) | 4
Cholestasis (Hepatobiliary disorders) | 3
Bronchitis (Infections and infestations) | 9
Gamma-glutamyltransferase increased (Investigations) | 4
Weight decreased (Investigations) | 3
Headache (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 6
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 7
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 6

LIMITATIONS AND CAVEATS:
Study treatment duration is at least 6 months for subjects with best achievable response after 3 months of treatment, of 9 months for subjects with best achievable response after 6 months of treatment and of 12 months in other cases.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.